CLINICAL TRIAL: NCT05080179
Title: The Interactive Effect of Social Norm and Self (vs. Others) Benefit Nudges on Downloads of COVID-19 Exposure Notification Smartphone Apps: A Randomized Trial
Brief Title: Impact of Nudges on Downloads of COVID-19 Exposure Notification Smartphone Apps: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 844564
Record Dates: First submitted 2021-10-12; First posted 2021-10-15 (Actual); Results first posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is a 2 (Self-Benefit vs. Other-Benefit) x 2 (Social Norm vs. No Social Norm) design. There are thus four conditions total.
Who Masked: Participant
Masking Description: Participants were unaware they were participating in a study, and were thus blinded to their treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Self-Benefit/Social Norm (Experimental): As part of their email, they read, "It can help you determine where and when to get testing, and how to get care if you need it." and "Over 650,000 Pennsylvanians have already downloaded the app!"
  Interventions: Behavioral: Self-Benefit/Social Norm
- Self-Benefit/No Social Norm (Experimental): As part of their email, they read, "It can help you determine where and when to get testing, and how to get care if you need it." They did not read any information about the number of Pennsylvanians who downloaded the app.
  Interventions: Behavioral: Self-Benefit/No Social Norm
- Other Benefit/Social Norm (Experimental): As part of their email, they read, "It can help you reduce your risk of unknowingly spreading the virus to your friends, family, and larger community." and "Over 650,000 Pennsylvanians have already downloaded the app!"
  Interventions: Behavioral: Other Benefit/Social Norm
- Other Benefit/No Social Norm (Experimental): As part of their email, they read, "It can help you reduce your risk of unknowingly spreading the virus to your friends, family, and larger community." They did not read any information about the number of Pennsylvanians who downloaded the app.
  Interventions: Behavioral: Other Benefit/No Social Norm

INTERVENTIONS:
Behavioral: Self-Benefit/Social Norm — As part of their email, they will read, "It can help you determine where and when to get testing, and how to get care if you need it." and "Over 650,000 Pennsylvanians have already downloaded the app!"
  Arms: Self-Benefit/Social Norm
Behavioral: Self-Benefit/No Social Norm — As part of their email, they will read, "It can help you determine where and when to get testing, and how to get care if you need it." They will not read any information about the number of Pennsylvanians who downloaded the app.
  Arms: Self-Benefit/No Social Norm
Behavioral: Other Benefit/Social Norm — As part of their email, they will read, "It can help you reduce your risk of unknowingly spreading the virus to your friends, family, and larger community." and "Over 650,000 Pennsylvanians have already downloaded the app!"
  Arms: Other Benefit/Social Norm
Behavioral: Other Benefit/No Social Norm — As part of their email, they will read, "It can help you reduce your risk of unknowingly spreading the virus to your friends, family, and larger community." They will not read any information about the number of Pennsylvanians who downloaded the app.
  Arms: Other Benefit/No Social Norm

SUMMARY:
Eligible participants who were active beneficiaries of a large insurer living in Pennsylvania were sent an email encouraging them to download the contact tracing app in Pennsylvania, COVID Alert PA.

Participants will be randomly assigned to one of four conditions in a 2 (Self-benefit vs. Other-Benefit) x 2 (Social Norms Present vs. Social Norms absent) design.

All participants received an email that said :

"COVID Alert PA is the official Exposure Notification App from the Pennsylvania Department of Health. Join Penn Medicine in the fight against COVID-19 and download COVID Alert PA today!"

---Investigators manipulated the content here---

"The app uses Bluetooth to sense when one person is in close contact with another person with the app. If someone tests positive for COVID-19, and they decide to upload the information to the health department, people who have the app and who have been in contact with them will be alerted.

If you are interested in downloading the app, please click COVID Alert PA. We appreciate you joining our efforts. Together we can beat COVID-19!"

In the Other-Benefit condition, it said: "It can help you reduce your risk of unknowingly spreading the virus to your friends, family, and larger community."

In the Self-Benefit condition, it said: "It can help you determine where and when to get testing, and how to get care if you need it."

In the Social Norms Present condition, it said: "Over 650,000 Pennsylvanians have already downloaded the app!"

In the Social Norms Absent condition, it said the statement about social norms above.

Participants who do not open the initial email received a follow-up email.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants were active beneficiaries of a large insurer living in Pennsylvania.

Exclusion Criteria:

* Participants who did not subscribe to offers and promotions emails were excluded, as were Medigap beneficiaries.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16903 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-01-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Independence Blue Cross (IBX), Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 39,938 Pennsylvania members of a larger insurer were randomly assigned to receive one email in a 2 (Focus on Self vs. Focus on Others) x 2 (Social Norm vs. No Social Norm) design. 16,903 members opened the e-mail - this is considered enrollment for the purposes of our study.
Pre-assignment Details: For this study, participants are considered enrolled once they open the e-mail that is sent to them by the large private insurer.
Period: Overall Study
Arm/Group | Self-Benefit/Social Norm | Self-Benefit/No Social Norm | Other Benefit/Social Norm | Other Benefit/No Social Norm
Started | 4232 | 4246 | 4211 | 4214
Completed | 353 | 380 | 355 | 744
Not Completed | 3879 | 3866 | 3856 | 3470

BASELINE CHARACTERISTICS:
Population: Pennsylvania members of a large private insurer.
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-Benefit/Social Norm | Self-Benefit/No Social Norm | Other Benefit/Social Norm | Other Benefit/No Social Norm | Total
Number analyzed (Participants) | 4232 | 4246 | 4211 | 4214 | 16903
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.85 (13.33) | 47.31 (13.26) | 46.74 (13.39) | 46.83 (13.43) | 46.93 (13.35)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 1720 | 1686 | 1762 | 1798 | 6966
  Female | 2512 | 2560 | 2449 | 2416 | 9937
  Unknown | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4232 | 4246 | 4211 | 4214 | 16903

OUTCOME MEASURES:

1. Primary Outcome: Click on Link to Download COVID Alert PA App
Description: The investigators measured choice to click on the link to download the COVID Alert PA app or not, conditional on opening the email. Because participants may not immediately open their e-mail, or may return to the e-mail to click the link, we allowed for a period of approximately 7 weeks or 48 days from date of initial e-mail for completion of outcome measure.
Time Frame: 48 days
Population: Pennsylvania members of large private insurer.
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Benefit/Social Norm | Self-Benefit/No Social Norm | Other Benefit/Social Norm | Other Benefit/No Social Norm
Number analyzed (Participants) | 4232 | 4246 | 4211 | 4214
Participants
  Number opened e-mail | 4232 | 4246 | 4211 | 4214
  Number clicked link | 353 | 380 | 355 | 744

ADVERSE EVENTS:
Time Frame: Study duration, 48 days
Description: No adverse events anticipated as study only involved sending e-mails and having people click links.
Arm/Group | Self-Benefit/Social Norm | Self-Benefit/No Social Norm | Other Benefit/Social Norm | Other Benefit/No Social Norm
All-Cause Mortality (participants affected / at risk) | 0/4232 | 0/4246 | 0/4211 | 0/4214
Serious Adverse Events (participants affected / at risk) | 0/4232 | 0/4246 | 0/4211 | 0/4214
Other Adverse Events (participants affected / at risk) | 0/4232 | 0/4246 | 0/4211 | 0/4214

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT05080179/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT05080179/SAP_001.pdf